CLINICAL TRIAL: NCT00786760
Title: Natural History of HPV Infection in Men: The HIM Study
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: MCC-13930; NCI CA098803-01a1 (Other: National Cancer Institute (NCI))
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Human Papillomavirus
Keywords: HPV; Papillomavirus; Infection; Sexually transmitted disease; STD
MeSH Terms: conditions — Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This study will create a specimen repository with which to test future novel hypotheses related to HPV infection among men. To assess other genetic, infectious, or environmental factors that may influence acquisition and persistence of HPV infections in men, whole blood, serum, exfoliated penile cell samples, and oral cells will be stored in aliquots for future analyses as funding becomes available. Using banked specimens preserved for DNA, RNA, and protein analyses, we will be able to assess novel biomarkers such as methylation status of oncogenic HPV, polymorphisms in genes involved in innate immunity (e.g., TLR genes), and mRNA of the E6 and E7 HPV oncoproteins in the future.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1. Men ages 18 - 44 years
  Interventions: Other: Cohort: 3000 men examined every 6 months for 4 years.
- 2. Men ages 45 - 70 years
  Interventions: Other: Pilot study: 150 men examined every 6 months for 4 years.

INTERVENTIONS:
Other: Cohort: 3000 men examined every 6 months for 4 years. — Prospectively assess HPV infection in a large cohort of men in the US , Mexico, and Brazil representing countries of low and high risk.
  Groups: 1. Men ages 18 - 44 years
Other: Pilot study: 150 men examined every 6 months for 4 years. — Prospectively assess HPV infection in a large cohort of men in the US , Mexico, and Brazil representing countries of low and high risk.
  Groups: 2. Men ages 45 - 70 years

SUMMARY:
The purpose of this study is to learn about the natural history of Human Papillomavirus (HPV) infection in men. The study will also find out what factors are linked to HPV in men including other sexually transmitted diseases (STDs). If participants test positive for syphilis, gonorrhea or chlamydia, we are required by law to report the results to the Florida Department of Health. Participants will be able to get free medical treatment from the Florida Department of Health for these STDs. Participants will be given a written report of the results of the STD testing.

DETAILED DESCRIPTION:
The study protocol will include a pre-enrollment run-in visit, a baseline visit (enrollment), and 8 additional visits after enrollment scheduled 6 months apart. Intervals of every 6 months were chosen to insure that both acquisition and loss of infections may be assessed, as studies in women indicate that median duration of oncogenic infections ranges between 7-9 months. Informed consent will occur during the run-in visit. The run-in and follow-up visits will include questionnaire administration, visual inspection of the skin and external genitalia, and the collection of urine, blood, oral cells, and penile skin samples If anogenital lesions are present at any of the clinic visits, they will be sampled as well.

ELIGIBILITY:
Inclusion Criteria:

* Men between 18 and 70 years of age, living in Southern Florida, US; Sao Paulo, Brazil; or state of Morelos, Mexico.
* Participant has never been told that they have penile or anal cancer or genital warts.
* Willing to attend scheduled visits every 6 months in the next 4 years.

Exclusion Criteria:

* Prospective participants with symptoms of any STD (excluding HPV) during screening will not be eligible to participate in the study until the STD (Sexually Transmitted Disease) infection is gone.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Men ages 18-44; a pilot study group, ages 45-70;
  2. residents of 3 sites - southern Florida, US, Sao Paulo, Brazil, or state of Morelos, Mexico
  3. report no prior diagnosis of penile or anal cancers
  4. have never been diagnosed with genital and anal warts
  5. have not participated in a HPV vaccine study
  6. report no prior diagnosis with acquired immune deficiency syndrome (AIDS) or human immunodeficiency virus (HIV)
  7. report no current penile discharge or burning during urination
  8. are not currently being treated for a sexually transmitted disease
  9. have not been imprisoned or homeless during the last 6 months
  10. have not been in drug treatment during the last 6 months
  11. no plan to relocate in the next 4 years
  12. willing to comply with 10 scheduled visits every 6 months for 4 years
Sampling Method: Probability Sample
Enrollment: 1431 (Actual)
Dates: Start 2005-06-14 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Cohort Selection | 3 years, 3 months
  The first specific aim is to establish the cohort of 3000 men ages 18 - 44 years who will be examined every 6 months for 4 years. To assess potential biases introduced by the run-in visit, Pearson's χ² test of association will be used to compare cohort participants and non-participants who attended the run-in visit with respect to known and potential HPV risk factors and HPV status. All analyses will be conducted using Intercooled STATA (StataCorp. 2001. Stata Statistical Software: Release 8.2 SE College Station, Texas: Stata Corporation).

SECONDARY OUTCOMES:
Incidence Rates of Specific HPV Type Infection | 4 years per participant
  The second specific aim is to determine the incidence and persistence of type-specific HPV infections. Estimates of the incidence rates of specific HPV type infection will be calculated on the basis of the number of cases in which a given type is detected for the first time in men who tested negative for that HPV type at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Giuliano, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute, Inc.
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Inc., Tampa, Florida, United States